CLINICAL TRIAL: NCT05796141
Title: Optimizing a Couples-Based mHealth Intervention for Weight Management
Brief Title: Becoming United in Lifestyle Decisions
Acronym: BUILD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Amy Gorin, Vice Provost for Health Sciences and Interdisciplinary Initiatives, University of Connecticut
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HR22-0023; 1R01DK132386-01 (NIH)
Record Dates: First submitted 2023-02-22; First posted 2023-04-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Overweight and Obesity
Keywords: couples; mobile weight loss treatment; weight control
MeSH Terms: conditions — Overweight; Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- Condition 1 (Experimental): 1) Core BWL Intervention
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention
- Condition 2 (Experimental): 1) Core BWL Intervention; 2) Home Environment Modifications
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Home Environment Modifications
- Condition 3 (Experimental): 1) Core BWL Intervention; 2) Autonomy Support Training
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Autonomy Support Training
- Condition 4 (Experimental): 1) Core BWL Intervention; 2) Autonomy Support Training; 3) Home Environment Modifications
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Autonomy Support Training; Behavioral: Home Environment Modifications
- Condition 5 (Experimental): 1) Core BWL Intervention; 2) Joint Feedback
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Joint Feedback
- Condition 6 (Experimental): 1) Core BWL Intervention; 2) Joint Feedback; 3) Home Environment Modifications
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Joint Feedback; Behavioral: Home Environment Modifications
- Condition 7 (Experimental): 1) Core BWL Intervention; 2) Joint Feedback; 3) Autonomy Support Training
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Joint Feedback; Behavioral: Autonomy Support Training
- Condition 8 (Experimental): 1) Core BWL Intervention; 2) Joint Feedback; 3) Autonomy Support Training; 4) Home Environment Modifications
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Joint Feedback; Behavioral: Autonomy Support Training; Behavioral: Home Environment Modifications
- Condition 9 (Experimental): 1) Core BWL Intervention; 2) Dyadic Action Planning
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Dyadic Action Planning
- Condition 10 (Experimental): 1) Core BWL Intervention; 2) Dyadic Action Planning; 3) Home Environment Modifications
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Dyadic Action Planning; Behavioral: Home Environment Modifications
- Condition 11 (Experimental): 1) Core BWL Intervention; 2) Dyadic Action Planning; 3) Autonomy Support Training
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Dyadic Action Planning; Behavioral: Autonomy Support Training
- Condition 12 (Experimental): 1) Core BWL Intervention; 2) Dyadic Action Planning; 3) Autonomy Support Training 4) Home Environment Modifications
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Dyadic Action Planning; Behavioral: Autonomy Support Training; Behavioral: Home Environment Modifications
- Condition 13 (Experimental): 1) Core BWL Intervention; 2) Dyadic Action Planning; 3) Joint Feedback
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Dyadic Action Planning; Behavioral: Joint Feedback
- Condition 14 (Experimental): 1) Core BWL Intervention; 2) Dyadic Action Planning; 3) Joint Feedback; 4) Home Environment Modifications
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Dyadic Action Planning; Behavioral: Joint Feedback; Behavioral: Home Environment Modifications
- Condition 15 (Experimental): 1) Core BWL Intervention; 2) Dyadic Action Planning; 3) Joint Feedback; 4) Autonomy Support Training
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Dyadic Action Planning; Behavioral: Joint Feedback; Behavioral: Autonomy Support Training
- Condition 16 (Experimental): 1) Core BWL Intervention; 2) Dyadic Action Planning; 3) Joint Feedback; 4) Autonomy Support Training; 5) Home Environment Modifications
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) intervention; Behavioral: Dyadic Action Planning; Behavioral: Joint Feedback; Behavioral: Autonomy Support Training; Behavioral: Home Environment Modifications

INTERVENTIONS:
Behavioral: Core Behavioral Weight Loss (BWL) intervention — Behavioral weight loss core (lessons, self weighing, self-monitoring, individual action planning, feedback and progress check ins)
Behavioral: Dyadic Action Planning — Participants will develop dyadic action plans together.
  Arms: Condition 10; Condition 11; Condition 12; Condition 13; Condition 14; Condition 15; Condition 16; Condition 9
Behavioral: Joint Feedback — Participants will see data on their partner's progress, in addition to their own weight and behavioral data.
  Arms: Condition 13; Condition 14; Condition 15; Condition 16; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Autonomy Support Training — Participants will receive training in how to create an autonomy supportive environment within their marriage/partnership.
  Arms: Condition 11; Condition 12; Condition 15; Condition 16; Condition 3; Condition 4; Condition 7; Condition 8
Behavioral: Home Environment Modifications — Participants will be trained in how to structure their home environment to support health behavior.
  Arms: Condition 10; Condition 12; Condition 14; Condition 16; Condition 2; Condition 4; Condition 6; Condition 8

SUMMARY:
The goal of this project is to investigate how to enhance the effects of an online-only (mHealth) couples weight loss program. This study will use an innovative methodological framework, the Multiphase Optimization Strategy (MOST), to test four different strategies for weight loss and partner support in addition to a core intervention (i.e., dyadic action planning, joint feedback on goal progress, autonomy support training, and home environment modifications).

ELIGIBILITY:
Inclusion Criteria:

* Married/cohabitating couple - both partners must be eligible
* BMI between 25-55kg/m2
* English speaking/reading
* Have a smartphone and reliable internet access
* Have active email address
* Willing to videoconference

Exclusion Criteria:

* Report being unable to walk 2 blocks without stopping
* Are currently participating in weight loss treatment, have a history of bariatric surgery, or lost ≥5% in the past 6-months
* Are pregnant or plan to become pregnant during the study period
* Report chest pain or loss of consciousness on the Physical Activity Readiness Questionnaire
* Report a medical condition that could jeopardize their safety in a weight control program with diet and exercise guidelines
* Report conditions that, in the judgment of the PI, would render them unlikely to follow the protocol (e.g. dementia)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Body Weight (kg) | Baseline to 6 months
  Weight change from baseline to 6 months. Weight will be objectively measured on a digital scale in the participant's home and weight change will be calculated.

SECONDARY OUTCOMES:
Goal Coordination (Wingrove Goal Coordination Scale) | Baseline, 3 months, 6 months
  Goal coordination (the extent to which partners integrate and align their weight management goals) will be measured with the Wingrove Goal Coordination Scale at baseline, 3, and 6 months.
Transactive Density | Baseline, 3 months, 6 months
  Interdependence of partners will be measured with the Inclusion of Others in the Self Scale at baseline, 3, and 6 months.
Shared Goal Representation | Baseline, 3 months, 6 months
  The Important Others Questionnaire will be used to capture shared goal representation at baseline, 3, and 6 months.
Home Food Environment (Household Food Inventory) | Baseline, 3 months, 6 months
  The home food environment will be measured with the Household Food Inventory, administered at baseline, 3, and 6 months.
Home Exercise Environment (Exercise Environment Questionnaire) | Baseline, 3 months, 6 months
  The home exercise environment will be measured with the Exercise Environment Questionnaire, administered at baseline, 3, and 6 months.
Dietary Intake | Baseline, 3 months, 6 months
  Dietary intake will be assessed at baseline and 3 months as a hypothesized behavioral mediator and at 6 months as a secondary outcome measure.
Physical Activity (Paffenbarger Physical Activity Questionnaire) | Baseline, 3 months, 6 months
  Physical activity will be assessed using the Paffenbarger Physical Activity Questionnaire at baseline and 3 months as a hypothesized behavioral mediator and at 6 months as a secondary outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- UConn's Weight Management Research Group, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No